CLINICAL TRIAL: NCT03501355
Title: Effects of Inspiratory Muscle and Endurance Training on Exercise Capacity, Respiratory Muscle Strength and Endurance and Quality of Life in Heart Failure Patients With Pacemaker
Brief Title: Effects of Inspiratory Muscle and Endurance Training in Heart Failure Patients With Pacemaker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gazi University 7
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Pacemaker
Keywords: pacemaker; inspiratory muscle training; exercise capacity; Quality of Life; Respiratory Muscle Strength

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training group (Active Comparator): Intervention:Inspiratory muscle strength training group received inspiratory muscle training (IMT) using POWERbreathe Classic threshold loading device
  Interventions: Device: Inspiratory muscle strength training
- Endurance training group (Active Comparator): Intervention: Inspiratory muscle endurance training group received inspiratory muscle endurance training (IMT) using POWERbreathe Classic threshold loading device
  Interventions: Device: Inspiratory muscle endurance training

INTERVENTIONS:
Device: Inspiratory muscle strength training — Treatment group will receive inspiratory muscle training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 50% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 50% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Arms: Strength training group
Device: Inspiratory muscle endurance training — Treatment group II will receive inspiratory muscle endurance training (IMT) using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 30% of maximal inspiratory pressure (MIP).
  The MIP will be measured at supervised session each week, and 30% of measured MIP value will be the new training workload.
  The treatment group will train for 30 min-per/day, 7 days/week, for 8 weeks. Six sessions at home and 1 session will be performed at department.
  Arms: Endurance training group

SUMMARY:
It is well-known that not only peripheral muscles, but also respiratory muscles muscle weakness and deconditioning play an important role in low exercise capacity of patients with Heart Failure (HF). Exercise training has been shown to improve exercise tolerance and quality of life in patients with heart disease. However, hearth failure patients with pacemaker such as implantable cardioverter defibrillators (ICDs), cardiac resynchronization pacemakers or defibrillators (CRT-P or CRT-D) have additional specific issues when performing exercise. No study investigated the effects of different inspiratory muscle training protocols. For this reason, we aimed to investigate the effects of inspiratory muscle training on outcomes in hearth failure patients with pacemaker

DETAILED DESCRIPTION:
Heart failure patients with pacemaker will be included. Primary outcome measurement is respiratory muscle strength, secondary outcomes are functional exercise capacity, peripheral muscle strength, pulmonary functions, maximal exercise capacity, fatigue, quality of life, depression, physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with Pacemaker who are clinically stable
* After 12 weeks of pacemaker implantation
* No change in medications over one month

Exclusion Criteria:

Patients with

* Severe cognitive disorders
* Pulmonary, neurological and orthopedic diseases
* Pregnant and lactating patients
* Acute infection or exacerbation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Maximal Exercise capacity | First day
  Incremental Shuttle Walk Test

SECONDARY OUTCOMES:
Inspiratory and expiratory muscle strength (MIP, MEP) | First day
  Mouth pressure device
Peripheral muscle strength | First day
  Hand held dynamometer
Pulmonary functions | First day
  Spirometry
Fatigue | Second day
  Fatigue Severity Scale (FSS) (Turkish version of scale) Patient choose a number from 1 to 7 that indicates how much the patient agrees with each statement, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 4 or higher generally indicates severe fatigue
Quality of life | Second day
  Short Form (SF-36) Health Survey (Turkish version of scale) The SF-36 is a 36 item questionnaire that measures eight multi-item dimensions of health: physical functioning (10 items) social functioning (2 items) role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items), and general health perception (5 items). For each dimension item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
Depression | Second day
  Montgomery Asberg Depression Rating Scale (MADRS) (Turkish version of scale) This assessment tool contains 10 items with a score from 0 to 6, thus the maximum score is 60. A higher score indicates a more severe depression.
Physical activity | Second day
  International Physical Activity Questionnaire (IPAQ) - Short Form (Turkish version of scale ) This questionnaire assesses, in minutes, the physical activity performed by the volunteers during the period of one week. The IPAQ considered all activities carried out by the volunteer (e.g. leisure, sport, exercise, and activities at home or in the garden). According to the responses, the volunteer is considered very active, active, irregularly active or sedentary, according to the intensity and time of the exercises practiced over the last week.
Health-related quality of life | Second day
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) (Turkish version of scale) 21 items rated on six-point Likert scales, representing different degrees of impact of HF on Heart Related Quality of Life (HRQoL), from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25).
Cognitive function | First day
  Mini mental state examination (MMSE)(Turkish version of scale ) The scale has a maximum score of 30 points. The questions have been grouped into seven categories, each rationally representing a different cognitive domain or function: Orientation to time (5 points); Orientation to place (5 points); Registration of three words (3 points); Attention and Calculation (5 points); Recall of three words (3 points); Language (8 points) and Visual Construction (1 point). The severity of cognitive impairment is classified as normal (30-27) mild cognitive impairment (26-20); moderate cognitive impairment (19-10); and severe cognitive impairment(< 10).
Functional exercise capacity | Second day
  6 minute walking test

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak-Güçlü, PhD, Study Director — Gazi University Faculty of Health Science Department of Physical Therapy and Rehabilitation; Nihan Katayıfçı, MSc, Study Chair — Mustafa Kemal University School of Physical Therapy and Rehabilitation; Fatih Şen, PhD, Principal Investigator — Mustafa Kemal University
Locations (1):
- Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alswyan AH, Liberato ACS, Dougherty CM. A Systematic Review of Exercise Training in Patients With Cardiac Implantable Devices. J Cardiopulm Rehabil Prev. 2018 Mar;38(2):70-84. doi: 10.1097/HCR.0000000000000289. PMID 29465496
- [Background] Belardinelli R, Capestro F, Misiani A, Scipione P, Georgiou D. Moderate exercise training improves functional capacity, quality of life, and endothelium-dependent vasodilation in chronic heart failure patients with implantable cardioverter defibrillators and cardiac resynchronization therapy. Eur J Cardiovasc Prev Rehabil. 2006 Oct;13(5):818-25. doi: 10.1097/01.hjr.0000230104.93771.7d. PMID 17001224
- [Background] Dougherty CM, Glenny RW, Burr RL, Flo GL, Kudenchuk PJ. Prospective randomized trial of moderately strenuous aerobic exercise after an implantable cardioverter defibrillator. Circulation. 2015 May 26;131(21):1835-42. doi: 10.1161/CIRCULATIONAHA.114.014444. Epub 2015 Mar 19. PMID 25792557
- [Background] Isaksen K, Munk PS, Giske R, Larsen AI. Effects of aerobic interval training on measures of anxiety, depression and quality of life in patients with ischaemic heart failure and an implantable cardioverter defibrillator: A prospective non-randomized trial. J Rehabil Med. 2016 Mar;48(3):300-6. doi: 10.2340/16501977-2043. PMID 26667151
- [Derived] Katayifci N, Bosnak Guclu M, Sen F. A comparison of the effects of inspiratory muscle strength and endurance training on exercise capacity, respiratory muscle strength and endurance, and quality of life in pacemaker patients with heart failure: A randomized study. Heart Lung. 2022 Sep-Oct;55:49-58. doi: 10.1016/j.hrtlng.2022.04.006. Epub 2022 Apr 23. PMID 35472660